CLINICAL TRIAL: NCT02910778
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Effect of Atorvastatin Treatment for 14 Days in Combination With an Acute Dose of Ticagrelor on Ischemia Reperfusion Induced Endothelial Dysfunction of the Forearm Vasculature in Healthy Male Subjects
Brief Title: The Effect of Ticagrelor With or Without Atorvastatin on Endothelial Function in Healthy Males
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wolzt, Prof. MD, Prof. MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FBF-Statin-Tica
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia | interventions — Atorvastatin; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): 80 mg atorvastatin for 14 days with a loading dose of 180 mg ticagrelor on day 15
  Interventions: Drug: Atorvastatin; Drug: Ticagrelor
- Placebo (Placebo Comparator): Placebo for 14 days with a loading dose of 180 mg ticagrelor on day 15
  Interventions: Drug: Placebo; Drug: Ticagrelor

INTERVENTIONS:
Drug: Atorvastatin — Subjects will receive 80 mg atorvastatin once daily for 14 days (until study day 15). On study day 15, 80 mg atorvastatin in combination with a loading dose of 180 mg ticagrelor will be administered.
  Arms: Atorvastatin
Drug: Placebo — Subjects will receive placebo once daily for 14 days (until study day 15). On study day 15, placebo in combination with a loading dose of 180 mg ticagrelor will be administered.
  Arms: Placebo
Drug: Ticagrelor

SUMMARY:
To test the effect of atorvastatin or placebo in combination with ticagrelor on ACh-induced vasodilatation of the forearm resistance vasculature as assessed by forearm blood flow (FBF) measurement before and 10 min after a 20 min forearm ischemia. The area under the dose-effect curve (AUC) of different ACh doses will be calculated and compared between treatment groups (atorvastatin + ticagrelor vs. placebo + ticagrelor) and different time points (pre-ischemia vs. post-ischemia).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects; 18 - 40 years of age
* Body mass index between 18 and 27 kg/m2
* Written informed consent
* Normal findings in medical & bleeding history
* Non-smoking

Exclusion Criteria:

* Regular intake of any medication including OTC drugs and herbals within 2 weeks before IMP administration
* Known coagulation disorders (e.g. haemophilia, von Willebrand´s disease)
* Known disorders with increased bleeding risk (e.g. peridontosis, haemorrhoids, acute gastritis, peptic ulcer, intestinal ulcer)
* Known sensitivity to common causes of bleeding (e.g. nasal)
* History of thromboembolism
* History of occlusive vascular diseases
* History of vascular anomalies
* History of hypercholesterolemia
* History of myopathy
* Impaired liver function (AST, ALT, gGT, bilirubin > 3 x ULN)
* Impaired renal function (serum creatinine > 1.3 mg/dl)
* Elevated creatinine-kinase or serum-myoglobin (> 3 x ULN)
* Any other relevant deviation from the normal range in clinical chemistry, haematology or urine analysis
* HIV-1/2-Ab, HbsAg or HCV-Ab positive serology
* Systolic blood pressure above 145 mmHg, diastolic blood pressure above 95 mmHg
* Known allergy against any test agent under study
* Regular daily consumption of more than on litre of xanthine-containing beverages or more than 40g alcohol
* Participation in another clinical trial during the preceding 3 weeks

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of Forearm blood flow (FBF) measurements of Acetylcholine (ACh) induced vasodilatation | Change of the AUC before and 10 min after forearm ischemia
  To test the effect of atorvastatin or placebo in combination with ticagrelor on ACh-induced vasodilatation of the forearm resistance vasculature as assessed by FBF measurement before and 10 min after a 20 min forearm ischemia

SECONDARY OUTCOMES:
Area under the curve (AUC) of Forearm blood flow (FBF) measurements of Glyceryltrinitrate (GTN) induced vasodilatation | Change of the AUC before and 10 min after forearm ischemia
  To test the effect of atorvastatin or placebo in combination with ticagrelor on GTN-induced vasodilatation of the forearm resistance vasculature as assessed by FBF measurement before and 10 min after a 20 min forearm ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weisshaar S, Litschauer B, Kerbel T, Wolzt M. Atorvastatin combined with ticagrelor prevent ischemia-reperfusion induced vascular endothelial dysfunction in healthy young males - A randomized, placebo-controlled, double-blinded study. Int J Cardiol. 2018 Mar 15;255:1-7. doi: 10.1016/j.ijcard.2017.12.067. Epub 2017 Dec 24. PMID 29288055